CLINICAL TRIAL: NCT02801890
Title: Autologous AD-MSC Transplantation in Peritoneal Dialysis Patients With Ultra Filtration Failure and Evaluation of Cellular and Molecular Effects of Mesenchymal Stem Cell Infusion on Peritoneal Fibrosis
Brief Title: Evaluation of Autologous Adipose Derived Mesenchymal Stromal Cells (AD-MSC) Transplantation in Ultra Filtration Failure (UFF)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-kidney-006
Record Dates: First submitted 2016-06-12; First posted 2016-06-16 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2016-12

CONDITIONS: Ultra Filtration Failure
MeSH Terms: interventions — Injections, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AD-MSC (Experimental): The patients with ultra filtration failure (UFF) underwent AD-MSC injection.
  Interventions: Biological: Intravenous injection
- Placebo (Placebo Comparator): The patients with ultra filtration failure (UFF) underwent Placebo injection.
  Interventions: Biological: Intravenous injection

INTERVENTIONS:
Biological: Intravenous injection — Intravenous injection of stem cell or placebo to the patients with The patients with ultra filtration failure (UFF) .

SUMMARY:
Peritoneal fibrosis may be occurred as a serious complication of peritoneal dialysis. It's the main factor of UFF that could lead to the Encapsulating Peritoneal Sclerosis (EPS). Using the potential features of MSCs in the treatment of fibrosis may offer new insights into reconstruction the damaged tissues. The project intends to transplant autologous MSCs to ten peritoneal dialysis patients with ultra-filtration failure. It's going to study infusion effects in clinical, cellular and molecular levels.

So in this trial, we will evaluate the effects of this intervention after intravenous injection of autologous adipose derived mesenchymal stem cells in 10 peritoneal dialysis patients with ultra filtration failure (UFF). Fifteen UFF patients are also considered as the control group. Then they will be followed 20, 45 and 90 days, and also 4 and 6 months after first injection.

DETAILED DESCRIPTION:
Chronic kidney disease is defined as a reduced glomerular filtration rate, increased urinary albumin excretion, or both, and is an increasing public health issue. Prevalence is estimated to be 8-16% worldwide. Stage 5 CKD is often called end-stage kidney disease and usually means that the patient requires renal replacement therapy (RRT), which may involve a kidney transplant or a form of dialysis. One of the options in RRT is continuous ambulatory peritoneal dialysis (CAPD). CAPD is characterized by a continuous removal of extracellular fluid by peritoneal membrane. It should be noted that like any other peritoneal dialysis therapy, CAPD has Short or long-term complications and UFF is the most common functional disorder in which the peritoneal ultrafiltration membrane damaged.

This project intends to evaluate, the role of autologous mesenchymal stem cells in improvement of peritoneal membrane function in peritoneal dialysis patients who have ultrafiltration failure up to 6 months.

In this study, 10 male and female subjects who are on peritoneal dialysis for at least two years and have ultrafiltration failure with age range of 18 to 70 years will be enrolled. Patients will be selected from peritoneal dialysis patients attending the peritoneal dialysis ward of Dr. Shariati hospital. The main inclusion criteria is to be on peritoneal dialysis for at least last two years and having Ultrafiltration failure. After obtaining the consent form, a sample of fat tissue will be obtained by a general surgeon under sterilized condition from patients and then in the specialized lab, the mesenchymal stem cells will be separated and cultured to reach appropriate numbers (106/kg). The cells will be injected through peripheral vein in hospital setting. Patients will be followed-up (clinically and laboratory) at baseline and at week 3, week 6, month 3, month 4 and month 6. The clinical assessment and peritoneal function tests will be performed in each visit. Outcome measures: The main outcome measures that periodically will be assessed include: D/P cr, D/P urea, D0/D glucose, PET, KT/V urea, Glomerular filtration rate (GFR)

ELIGIBILITY:
Inclusion Criteria:

1. peritoneal dialysis for at least last two years and
2. Ultrafiltration failure
3. Both genders
4. Age 18-70 years
5. inform consent signing

Exclusion Criteria:

1. Inability of patients to attend visits and regular testing
2. Estimated lifetime less than one year
3. Use of immunosuppressive drugs
4. Pregnancy
5. Malignancy
6. Coagulative disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Systemic infection | 6months
  Evaluation the rate of systemic infection in patients with UFF after cell therapy.
Hepatic failure | 6 months
  Evaluation the rate of hepatic failure in patients with UFF after cell therapy.
Renal failure | 6 months
  Evaluation the rate of renal failure in patients with UFF after cell therapy.

SECONDARY OUTCOMES:
Ratio of 4-hour dialysate/plasma creatinine (D/P Cr). | 6 months
  Evaluation the change of (D/P Cr) in patients with UFF after cell therapy.
Ratio of 4-hour dialysate/plasma urea (D/P urea ) | 6 months
  Evaluation the change of D/P in patients with UFF after cell therapy.
Ratio of dialysate glucose concentrations (D/D glucose ) | 6 months
  Evaluation the change of D/D glucose in patients with UFF after cell therapy.
peritoneal membrane transport function | 6 months
  Assessment of peritoneal membrane transport function by peritoneal equilibration test (PET)
Glomerular filtration rate (GFR): | 6 months
  Evaluation the change of Glomerular filtration rate (GFR) in patients with UFF after cell therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Department of Regenerative Biomedicine at the Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.; Gholamreza Pourmand, MD, Study Director — Urology Research Center, Sina Hospital, Tehran University of Medical Sciences, Iran.; Iraj Najafi, MD, Study Director — Urology Research Center, Sina Hospital, Tehran University of Medical Sciences, Iran.; Sudabeh Alatab, MD, Principal Investigator — Sudabeh; Soroosh Shekarchian, MD, Principal Investigator — Department of Regenerative Biomedicine at the Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.; Reza Moghadasali, PhD, Principal Investigator — Department of Regenerative Biomedicine at the Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No